CLINICAL TRIAL: NCT02368717
Title: A Randomized, Double-blind, Placebo-controlled, Multi-centre, Superiority Study Investigating the Efficacy and Safety of PENTASA Enema Compared With Placebo Enema for 4-Week Treatment in Chinese Patients With Left-sided Active Ulcerative Colitis (UC) Followed by a Maximal 28-Week Open-Label Extension Phase of PENTASA Enema and/or PENTASA Tablets
Brief Title: An Efficacy and Safety Study of PENTASA in Chinese Patients With Left-sided Active Ulcerative Colitis Followed by a 24-Week Open-Label Extension Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000101
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalazine (Experimental): Mesalazine Enema
  Interventions: Drug: Mesalazine Enema
- Placebo (Placebo Comparator): Placebo Enema
  Interventions: Drug: Placebo Enema

INTERVENTIONS:
Drug: Mesalazine Enema
  Other Names: PENTASA® Enema
  Arms: Mesalazine
Drug: Placebo Enema
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of 4-week double-blind treatment with PENTASA enema compared with placebo enema in Chinese patients with mild to moderate active left-sided ulcerative colitis, followed by a maximal 28-week open-label extension phase with PENTASA enema and/or PENTASA tablets.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent mild to moderate left-sided active ulcerative colitis
* Mayo score of at least 4 but not greater than 10 points and a score of ≥ 2 for colonoscopy
* Extent of colonic involvement and endoscopy subscore of Mayo score as confirmed by colonoscopy
* The patient is compliant with Patient Daily Diary by having adequately responded to the questions on ≥5 of the most recent full 7 days before the Randomization Visit
* Negative stool test at screening to rule out parasites and bacterial pathogens

Exclusion Criteria:

* Patients receiving > 2g/day of oral 5-aminosalicylic acid (5-ASA) products, or receiving topical rectal 5-ASA > 3g/week, within 7 days prior to screening
* Severe/fulminant ulcerative colitis or toxic dilatation of the colon
* Prior bowel resection surgery
* Patients allergic to 5-ASA and derivative, any of the excipients, aspirin, or salicylates
* Patients with one or more of the diseases: bacillary dysentery, amebic dysentery, chronic schistosomiasis, intestinal tuberculosis and Crohn's disease
* Patients who are unable to fill in the Patient Daily Diary or follow data-capturing procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01-05 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Clinical remission after 4 weeks treatment | At week 4
  Defined as a total Mayo score ≤2 points, with no subscore >1 point

SECONDARY OUTCOMES:
Clinical response after 4 weeks treatment | At week 4
  Defined as a decrease from baseline in total Mayo score ≥3 points and ≥ 30 percent, with an accompanying decrease in the subscore for rectal bleeding ≥ 1 point or an absolute subscore for rectal bleeding of 0 or 1 point
Change in Quality of Life | From baseline to week 4
  Based on the Inflammatory Bowel Disease Questionnaire (IBDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- The 6th hospital affiliated to Zhongshan University (there may be other sites in this country), Guangzhou, China